CLINICAL TRIAL: NCT06518850
Title: A Multicentre Study of Clinical Features and Efficacy of Small Intestinal Bacterial Overgrowth in Abdominal Distension Patients
Brief Title: Study of Clinical Features and Efficacy of Small Intestinal Bacterial Overgrowth in Patients With Abdominal Distension
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Navy General Hospital, Beijing (Other); Air Force Military Medical University, China (Other); Beijing Tongren Hospital (Other); Beijing Friendship Hospital (Other); Beijing Chao Yang Hospital (Other); Beijing Tiantan Hospital (Other); The Luhe Teaching Hospital of the Capital Medical University (Other); China-Japan Friendship Hospital (Other); Beijing Aerospace General Hospital (Other); Beijing Jishuitan Hospital (Other); Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Jing-Nan Li, Chief physician, Professor, Peking Union Medical College Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: I-23PJ1228
Record Dates: First submitted 2024-07-13; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Small Intestine Bacterial Overgrowth
Keywords: small intestine bacterial overgrowth; oral cecum transit time; abdominal distention
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Comparator（Normal oral cecum transit time） (Sham Comparator): Normal oral cecum transit time +functional abdominal distention +small intestinal bacterial overgrowth.Rifaximin (0.2g/ time, 4 times/day) was discontinued after 14 days of treatment.
  Interventions: Drug: Rifaximin
- Experimental（Abnormal oral cecum transit time） (Experimental): Abnormal oral cecum transit time +functional abdominal distention +small intestinal bacterial overgrowth.Rifaximin (0.2g/ time, 4 times/day) was discontinued after 14 days of treatment.
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Both groups were treated with rifaximin for 14 days, during which follow-up records were reported by the subjects in the daily reference case report form. Methane and hydrogen breath tests were repeated 2 weeks after withdrawal.

SUMMARY:
Most studies of bloating have focused on functional factors, while data on organic abdominal distention are rare, and studies that combine small intestine bacterial overgrowth and/or oral cecum transit time abnormalities are more urgent to explore. On this basis, patients with functional abdominal distension complicated with small intestine bacterial overgrowth were divided according to whether there was abnormal oral cecum transit time, and given the same treatment plan. The relief effect of abdominal distension, small intestine bacterial overgrowth turning negative and oral cecum transit time recovery were observed, so as to further clarify the cause of abdominal distension patients.

DETAILED DESCRIPTION:
Part 1 Clinical characteristics of small intestinal bacterial overgrowth in patients with abdominal distension of different etiologies The clinical characteristics of small intestine bacterial overgrowth and oral cecum transit time in patients with abdominal distention of different etiology (organic and functional) were studied to lay a foundation for further exploration of treatment of functional abdominal distention.

Part 2 Efficacy observation of functional abdominal distention combined with small intestine bacterial overgrowth To observe the effect of antibiotics on abdominal distension in patients with functional abdominal distension complicated with small intestine bacterial overgrowth, and observe the effect of rifaximin on small intestine bacterial overgrowth and oral cecum transit time, so as to provide new ideas for the diagnosis and treatment of abdominal distension patients.

ELIGIBILITY:
Inclusion criteria:

Part 1 Clinical characteristics of small intestinal bacterial overgrowth in patients with abdominal distension of different etiologies

1. Age 18-60 years old and gender;
2. The chief complaint is abdominal distension and/or abdominal distension, abdominal distension and/or abdominal distension more prominent than other symptoms.

Part 2 Efficacy observation of functional abdominal distention combined with small intestine bacterial overgrowth

1. Patients with functional abdominal distension and small intestinal bacterial overgrowth were selected in Part 1;
2. No drug contraindications.

Exclusion criteria:

Part 1 Clinical characteristics of small intestinal bacterial overgrowth in patients with abdominal distension of different etiologies

1. Preparation for pregnancy, pregnancy, breastfeeding women, or overall poor compliance, or other conditions that the investigator believes need to be excluded;
2. History of malignant tumors, history of abdominal surgeries;
3. Food intolerance, confirmed or suspected lactose intolerance;
4. Diagnosis of urinary system (chronic kidney disease, etc.), immune system (scleroderma, etc.), nervous system (Parkinson's disease, etc.), mental system (depression, etc.) and other diseases outside the digestive system;
5. Antibiotics and microecological preparations should be used within two weeks. Use motility enhancers, secretagogues, antifoaming agents, spasmolytics, opioids, antidepressants and other medications within a week.

Part 2 Efficacy observation of functional abdominal distention combined with small intestine bacterial overgrowth

1. Antibiotics and microecological preparations should be used within two weeks;
2. Use motility enhancers, secretagogues, antifoaming agents, spasmolytics, opioids, antidepressants and other medications within a week.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Part 1 Positive rate of small intestinal bacterial overgrowth | 1 day
  Positive rate of small intestinal bacterial overgrowth in organic and functional abdominal distension
Part 1 Abnormal rate of oral cecum transit time | 1 day
  Abnormal rate of oral cecum transit time in organic and functional abdominal distension
Part 2 Effective rate of abdominal distension | 2 weeks
  Total effective rate (%) = Obvious effective rate (%) + Effective rate (%)
  1. Obvious effect: the degree and frequency of abdominal distension score improved, or even completely disappeared, small intestinal bacterial overgrowth negative
  2. Effective: the degree and frequency of abdominal distension score improved, small intestinal bacterial overgrowth positive
  3. Ineffective: the degree and frequency of abdominal distension score did not improve
Part 2 Negative conversion rate of small intestinal bacterial overgrowth and oral cecum transit time | 2 weeks
  1. Negative conversion rate of small intestinal bacterial overgrowth (%) =Number of small intestinal bacterial overgrowth negative after treatment/ Number of functional abdominal distention in Part 2*100%
  2. Negative conversion rate of oral cecum transit time (%) =Number of oral cecum transit time normal after treatment/ Number of experimental in Part 2*100%

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Nan Li, MD,Ph.D, Principal Investigator — Peking Union Medical College Hospital